CLINICAL TRIAL: NCT05346302
Title: Persistent Readiness Through Early Prediction Immunization Study
Acronym: PREP DOD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Philips Healthcare (Industry); US Department of Defense - Defense Threat Reduction Agency (Unknown)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PREP DOD
Record Dates: First submitted 2022-02-01; First posted 2022-04-26 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Response
Keywords: commercial off the shelf wearable devices; large-scale machine learning; biomarkers; early warning of infection; predictive model of illness severity; predictive model of recovery
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Vi polysaccharide vaccine, typhoid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled vaccine administration (pneumococcal (PPSV23), typhoid (inactivated), or saline)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pneumococcal (PPSV23) vaccine (Active Comparator): PNEUMOVAX 23 is a clear, colorless solution. Each 0.5-mL dose of vaccine contains 25 micrograms of each polysaccharide type in isotonic saline solution containing 0.25% phenol as a preservative under the supervision of a licensed pharmacist.
  Interventions: Drug: Pneumovax 23
- Typhoid (inactivated) vaccine (Active Comparator): Typhoid vaccine is a clear, colorless solution. Each dose of 0.5 mL is formulated to contain 25 mcg of purified Vi polysaccharide in a colorless isotonic phosphate buffered saline (pH 7 ± 0.3), 4.150 mg of Sodium Chloride, 0.065 mg of Disodium Phosphate, 0.023 mg of Monosodium Phosphate, and 0.5 mL of Sterile Water for Injection under the supervision of a licensed pharmacist.
  Interventions: Drug: Typhim VI
- Saline (Placebo Comparator): Saline will be purchased commercially and compounded under the supervision of a licensed pharmacist in sterile syringes for administration of the placebo group.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Pneumovax 23 — At +14 days from enrollment in the trial, participants will receive a vaccine administered via intramuscular route only.
  Arms: Pneumococcal (PPSV23) vaccine
Drug: Typhim VI — At +14 days from enrollment in the trial, participants will receive a vaccine administered via intramuscular route only.
  Arms: Typhoid (inactivated) vaccine
Other: Saline — At +14 days from enrollment in the trial, participants will receive a vaccine administered via intramuscular route only.
  Arms: Saline

SUMMARY:
This study will enroll volunteers in an open-format (outside hospital) setting, to complete novel data collection/analysis of biomarkers, facial images, and audio-recording to establish an optimal set of parameters to predict emergent cases of infection via an early warning score, along with actionable personalized information.

DETAILED DESCRIPTION:
The objective of the study is to collect data from participants for a period of 4 weeks. These data will be used for developing and testing an algorithm for early detection of infection.

At the end of week two, subjects will receive an immunization in a double-blind randomized placebo-controlled fashion. Vaccines to be administered will be pneumococcal (PPSV23), typhoid (inactivated), or saline. Administration of these vaccines often cause mild 'infection-like' inflammation response. Pneumococcal infection causes pneumonia and can lead to sepsis and the PPSV23 vaccination will induce mild symptoms related to the immune system activation including local reaction in 50% of the cases and fever and malaise in 1% of the cases. Typhoid fever is caused by salmonella Typhi bacteria and its effects can range from gastrointestinal symptoms to sepsis. Injectable typhoid vaccine (inactivated) side effects will induce mild symptoms related to the immune system activation and can include local reaction in 6% of the cases and fever, malaise, headache and sometimes diarrhea in 1% of the cases.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40 (inclusive)
* Subject is judged to be in satisfactory health based on medical history, physical examination
* Ability to walk, sit down and stand up independently
* Willingness and ability to comply with the protocol
* ownership and use of smartphone
* ownership and use of laptop

Exclusion Criteria:

* Subject has planned elective surgery requiring 2 or more days of hospitalization during the entire study
* Active dependence of alcohol or drugs (self-reported)
* Known allergy to any of the following:
* Components of the vaccine/placebo
* Diagnosed and active treatment of chronic disease:
* Diabetes (Type 1 or 2)
* Active malignancy
* Heart disease
* Kidney disease
* Liver disease
* HIV/AIDS
* Hepatitis A, B, or C
* Asthma (moderate to severe)
* (possible/desire to be) pregnancy (confirmed via urine pregnancy test)
* Subject is currently enrolled in a study with an investigational compound or device
* Subject has already received the pneumococcal (PPSV23) vaccine
* Subject has already received the typhoid (inactivated) vaccine
* Subject has received any other investigational vaccination within 4 weeks of enrollment
* Any other condition that interfere with the definition 'healthy" based on self-report and according to the PI/study physician's judgement based on medical history, use of medication, and physical exam.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Questionnaires, self-reported changes in general physical health, and physiological measurements to predict of type of vaccine administered | up to 4 weeks
  Using a daily electronic questionnaire to collect data that self-reporting changes in general physical health and physiological measurements to identify the type of intervention

SECONDARY OUTCOMES:
Electrocardiography Morphology | up to 4 weeks
  Comparison of signals from standard electrocardiography (ECG) and wearable devices measuring the time elapsed between features of the electrical activity of the heart (e.g., P-wave, PR interval, PR segment, QRS complex, QRS duration, ST segment, J point, TP interval, T-wave, U-wave, QT duration, QTc interval)
Heart Rate | up to 4 weeks
  Comparison of signals from standard electrocardiography (ECG) and wearable devices measuring beats per minute of the heart
Heart Rate Variability | up to 4 weeks
  Comparison of signals from standard electrocardiography (ECG) and wearable devices measuring variation in the time interval between consecutive heartbeats in milliseconds
Body Temperature | up to 4 weeks
  Comparison of signals from contact infrared forehead thermometer and wearable devices measuring body surface temperature
Blood pressure (systolic and diastolic) | up to 4 weeks
  Comparison of signals from standard upper arm cuff and wearable devices measuring bloodpressure
Respiratory Rate | up to 4 weeks
  Comparison of signals from nasal cannula and wearable devices measuring number of breaths per minute
Amount of End-tidal Carbon Dioxide | up to 4 weeks
  Collection from nasal cannula to measure amount of EtCO2 in exhaled breath
Oxygen Saturation | up to 4 weeks
  Comparison of signals from fingertip pulse oximeter and wearable devices measuring level of oxygen saturation in blood
Assessment of the type and relative abundance of protein and lipids contained in Exhaled Breath Condensate | at enrollment, and +7, +14, +16, +21, +28 days of enrollment
  Measurement of presence and amount of components (e.g., protein, lipids) in exhaled breath condensate as determined by liquid chromatography tandem chromatography mass spectrometry
Assessment of the type and relative abundance of Volatile Organic Compounds contained in exhaled breath | at enrollment, and +7, +14, +16, +21, +28 days of enrollment
  Measurement of presence and amount of volatile organic compounds (e.g., ethanol, acetone, etc) in breath by comprehensive gas chromatography mass spectrometry (GCxGC-MS)
Digital photo of the face to assess changes in general facial features | up to 4 weeks
  Comparison of facial features taken with on-site digital camera and mobile device to compare general facial features such as 2-D facial landmarks, 3-D head pose, Deeply embedded facial expression features, and facial expressions via tools like Mediapipe face mesh or deepface and skin tone histograms at [RGB, HSV and YCbCr]
Digital photo of the face to assess changes in eyes | up to 4 weeks
  Comparison of facial features taken with on-site digital camera and mobile device to compare general features of the eye such as 2-D eyes and iris landmarks and shapes, Gaze directions of two eyes, Pixel histograms of Iris, pupil, and sclera at [RGB, HSV and YCbCr], Deeply embedded iris recognition features (via tools like irisRecognition), or eye texture features (Gabor filter banks, Haralick features) using tools like Mediapipe Iris
Digital photo of the face to assess changes in other facial components | up to 4 weeks
  Comparison of facial features taken with on-site digital camera and mobile device to compare general features Pixel histograms of: nose, forehead, left cheek, right cheek, mouth and lips at [RGB, HSV and YCbCr] using part segmentation done with Mediapipe facemesh
Digital audio recording of vocal expressions to assess changes in vowel components | up to 4 weeks
  Comparison of vocal features taken with on-site digital microphone and mobile device to compare vowel components of: mean frequency (Hz), variation coefficient (%), jitter factor (%), mean intensity (dB), shimmer factor (%), and noise to harmony ratio (dB).
Digital audio recording of vocal expressions to assess frequency changes in speech prosody components | up to 4 weeks
  Comparison of vocal features taken with on-site digital microphone and mobile device to compare speech prosody components of: mean frequency (Hz), minimal frequency (Hz), maximal frequency (Hz), dynamic (Hz).
Digital audio recording of vocal expressions to assess variation changes in speech prosody components | up to 4 weeks
  Comparison of vocal features taken with on-site digital microphone and mobile device to compare speech prosody components of: median frequency variation coefficient (%), percentage of pauses (%), percentage of pauses within words (%), fragmentation of vowels (%), and stop-consonant spirantization (%).
Digital audio recording of vocal expressions to assess time domain changes in speech prosody components | up to 4 weeks
  Comparison of vocal features taken with on-site digital microphone and mobile device to compare speech prosody components of: mean duration of speech between two pauses (seconds), total amount of syllables (syllables/s), total amount of pure speech (syllables/s), articulation rate (syllables/s), time between pauses (s), SPIR index of rhythmicity (words/min), voice onset time (s).
Continuous Glucose Monitoring | up to 2 weeks
  Using the DexCom G6 continuous glucose monitoring will be done for the week prior to and following the vaccination
Changes in physical health as measured by the Medical Symptoms Questionnaire (MSQ) | +7, +14, +16, +21, +28 days of enrollment
  The MSQ is administered by study staff for self-reporting of presence and severity of changes in symptoms in body symptoms: digestive tract, ears, emotions, energy/activity, eyes, head, heart, joint/muscles, lungs, mind, mouth/throat, nose, skin, weight, other.
Changes in gut function as measured by Gastrointestinal Symptom Rating Scale (GSRS) | +7, +14, +16, +21, +28 days of enrollment
  The GSRS is self-administered questionnaire regarding gut function and associated symptoms. It is composed of 15 items (7-Point Likert Scale) assessing Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Scores range from 15 to 105 with a higher score indicating more discomfort.
Changes in physical activity as measured by the short International Physical Activity Questionnaire (IPAQ) | +7, +14, +21, +28 days of enrollment
  The IPAQ is a self-administered questionnaire to provide a set of well-developed instruments that can be used internationally to obtain comparable estimates of physical activity.
Changes in daily dietary intake as measure by the Food Frequency Questionnaire (FFQ) | +7, +28 days of enrollment
  The FFQ is a self-administered questionnaire to provide an estimation of dietary protein intake.
Changes in duration and quality of sleep as measured by Pittsburgh Sleep Quality Index (PSQI) | +7, +28 days of enrollment
  The PSQI is a self-administered questionnaire to assesses sleep quality and disturbances. 19 individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Changes in physical activity as measured by the Baecke Physical Activity Questionnaire | +7, +28 days of enrollment
  Self-administered, 16-item questionnaire measuring physical activities in 3 categories: occupational, sport, recreational/leisure
Changes in quality of life as measured by Short Form (SF) Health Survey (SF36) | +7, +28 days of enrollment
  Self administered questionnaire that measures each of the following eight health concepts: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); Mental Health (MH) as well as a reported Health Transition item (HT)
Renal function panel Albumin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Albumin
Renal function panel BUN/Creatinine Ratio | +14, +16, +21 days of enrollment
  Blood sample taken to measure BUN/Creatinine Ratio (calculated)
Renal function panel Calcium | +14, +16, +21 days of enrollment
  Blood sample taken to measure Calcium
Renal function panel Carbon Dioxide | +14, +16, +21 days of enrollment
  Blood sample taken to measure Carbon Dioxide
Renal function panel Chloride | +14, +16, +21 days of enrollment
  Blood sample taken to measure Chloride
Renal function panel Creatinine | +14, +16, +21 days of enrollment
  Blood sample taken to measure Creatinine
Renal function panel Estimated Glomerular Filtration Rate | +14, +16, +21 days of enrollment
  Blood sample taken to measure Estimated Glomerular Filtration Rate (calculated)
Renal function panel Glucose | +14, +16, +21 days of enrollment
  Blood sample taken to measure Glucose
Renal function panel Phosphate | +14, +16, +21 days of enrollment
  Blood sample taken to measure Phosphate (as Phosphorus)
Renal function panel Potassium | +14, +16, +21 days of enrollment
  Blood sample taken to measure Potassium
Renal function panel Sodium | +14, +16, +21 days of enrollment
  Blood sample taken to measure Sodium
Renal function panel Urea Nitrogen | +14, +16, +21 days of enrollment
  Blood sample taken to measure Urea Nitrogen
Hepatic function panel Total Protein | +14, +16, +21 days of enrollment
  Blood sample taken to measure Total Protein
Hepatic function panel Albumin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Albumin
Hepatic function panel Globulin (calculated) | +14, +16, +21 days of enrollment
  Blood sample taken to measure Globulin (calculated)
Hepatic function panel Albumin/Globulin Ratio | +14, +16, +21 days of enrollment
  Blood sample taken to measure Albumin/Globulin Ratio (calculated)
Hepatic function panel Total Bilirubin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Total Bilirubin
Hepatic function panel Direct Bilirubin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Direct Bilirubin
Hepatic function panel Indirect Bilirubin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Indirect Bilirubin (calculated)
Hepatic function panel Alkaline Phosphatase | +14, +16, +21 days of enrollment
  Blood sample taken to measure Alkaline Phosphatase
Hepatic function panel Aspartate transaminase | +14, +16, +21 days of enrollment
  Blood sample taken to measure Aspartate transaminase
Hepatic function panel Alanine Aminotransferase | +14, +16, +21 days of enrollment
  Blood sample taken to measure Alanine Aminotransferase
Lipid panel | +14, +16, +21 days of enrollment
  Blood sample taken to measure Total Cholesterol, HDL Cholesterol, LDL Cholesterol, Triglycerides, VLDL Cholesterol
CBC (DIFF/PLT) White blood cell count | +14, +16, +21 days of enrollment
  Blood sample taken to measure White blood cell count
CBC (DIFF/PLT) red blood cell count | +14, +16, +21 days of enrollment
  Blood sample taken to measure red blood cell count
CBC (DIFF/PLT) Hemoglobin | +14, +16, +21 days of enrollment
  Blood sample taken to measure Hemoglobin
CBC (DIFF/PLT) Hematocrit | +14, +16, +21 days of enrollment
  Blood sample taken to measure Hematocrit
CBC (DIFF/PLT) mean corpuscular volume | +14, +16, +21 days of enrollment
  Blood sample taken to measure mean corpuscular volume
CBC (DIFF/PLT) mean corpuscular hemoglobin | +14, +16, +21 days of enrollment
  Blood sample taken to measure mean corpuscular hemoglobin
CBC (DIFF/PLT) corpuscular hemoglobin concentration | +14, +16, +21 days of enrollment
  Blood sample taken to measure mean corpuscular hemoglobin concentration
CBC (DIFF/PLT) red cell distribution width | +14, +16, +21 days of enrollment
  Blood sample taken to measure red cell distribution width
CBC (DIFF/PLT) Platelet Count | +14, +16, +21 days of enrollment
  Blood sample taken to measure Platelet Count
CBC (DIFF/PLT) mean platelet volume | +14, +16, +21 days of enrollment
  Blood sample taken to measure mean platelet volume
CBC (DIFF/PLT) Differential | +14, +16, +21 days of enrollment
  Blood sample taken to measure Differential (Absolute and Percent - Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils)
Highly Sensitive CRP | +14, +16, +21 days of enrollment
  Blood sample taken to measure Highly Sensitive C-Reactive Protein
Hemoglobin A1C | +14 days of enrollment
  Blood sample taken to measure hemoglobin A1C
Body Composition using Dual Energy X-Ray Absorptiometry bone density | at enrollment
  Measurement of bone mineral density (g/cm^2)
Body Composition using Dual Energy X-Ray Absorptiometry Muscle | at enrollment
  Measurement of muscle mass (kg)
Body Composition using Dual Energy X-Ray Absorptiometry Fat | at enrollment
  Measurement of fat mass (kg)
Measurement of daily physical activity using accelerometry sensors | up to 4 weeks
  Changes in physical activity detected by accelerometry data of wearable devices

OTHER OUTCOMES:
Development of personalized algorithm to provide an estimate of probability of onset of infection using activity and physiological measures | through study completion, up to 4 weeks
  Apply machine learning algorithms to data collected from clinical setting and wearable devices at various time scales relative to symptoms that are represented by percent score between 0-100%.
Development of personalized algorithm to provide an estimated index of severity of infection using activity and physiological measures | through study completion, up to 4 weeks
  Apply machine learning algorithms to data collected from clinical setting and wearable devices at various time scales relative to symptoms to estimate the acuity/intensity of care associated with infection ranging from 0-10.
Development of personalized algorithm to provide an estimated score related to time until recovery of infection using activity and physiological measures | through study completion, up to 4 weeks
  Apply machine learning algorithms to data collected from clinical setting and wearable devices at various time scales relative to symptoms to be reported in hours.
Development of personalized algorithm to provide detect the systems involved (respiratory vs gastrointestinal vs other) in infection using activity and physiological measures | through study completion, up to 4 weeks
  Apply machine learning algorithms to data collected from clinical setting and wearable devices at various time scales relative to symptoms to generate a probability score of systems involved in infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University - CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schrader SE, Hansen JR, O'Bryon I, Ruebush LE, Deutz NE, Wahl JH, Deatherage Kaiser BL. Volatile organic compound and proteomics data from the same exhaled breath condensate sample. J Breath Res. 2025 Aug 4;19(4). doi: 10.1088/1752-7163/adf34d. PMID 40701160
- [Derived] Wang C, Damiano RJ, Ruebush LE, Engelen MPKJ, Mariani S, Liu L, Silva I, Borhani S, Cote GL, Conroy B, McFarlane D, Deutz NEP. A randomized, triple-blinded, placebo-controlled clinical trial evaluating immune responses of Typhim Vi and PPSV23 vaccines in healthy adults: The PREP study. Vaccine. 2024 Dec 2;42(26):126292. doi: 10.1016/j.vaccine.2024.126292. Epub 2024 Sep 7. PMID 39245584